CLINICAL TRIAL: NCT05496296
Title: Randomized, Controlled, Open-Label, Parallel Group, Multi-Center, Prospective Phase 4 Study Comparing the Efficacy of Transforming Powder Dressing to NPIAP Recommended Standard of Care Therapies in Stage 2, 3 and 4 Pressure Injuries
Brief Title: Comparison of Transforming Powder Dressing to NPIAP Recommended Standard of Care Therapies in Stage 2, 3 and 4 Pressure Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ULURU Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: U-C-TPD-2022-01
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pressure Ulcers Stage II; Pressure Ulcers Stage III; Pressure Ulcer, Stage IV
Keywords: Wound care; Quality of life; Pain
MeSH Terms: conditions — Pressure Ulcer; Pain

STUDY DESIGN:
Intervention Model Description: Randomized, Prospective, Controlled, Open-label, Parallel Group, Multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care Dressing for Pressure Injury (Active Comparator): Standard wound dressings recommended by the National Pressure Injury Advisory Panel (NPIAP), according to the wound stage, will be utilized to treat pressure injuries. These include hydrocolloid, hydrogel, polymeric membranes, foam, collagen dressings, and negative pressure wound therapy. Dressings will be changed according to wound conditions, and type of dressing selected.
  Interventions: Device: Altrazeal® Transforming Powder Dressing
- Altrazeal® Transforming Powder Dressing (Active Comparator): Altrazeal® Transforming Powder Dressing will be applied during the Baseline visit. It should be left in place for up to 30 days, and topped off (additional powder applied if needed) at each subsequent visit. Secondary dressing, including a contact layer over the Altrazeal® and a secondary dressing (like gauze or foam) may be applied over the contact layer.
  Interventions: Device: Altrazeal® Transforming Powder Dressing

INTERVENTIONS:
Device: Altrazeal® Transforming Powder Dressing — Pressure injury wounds will be evaluated at each study visit (cleaned, photographed, measured) and a dressing will be applied according to the study arm
  Other Names: Standard of Care wound dressings (such as foam, hydrocolloid, collagen, etc)

SUMMARY:
Pressure injuries, commonly known as pressure ulcers, affect over 2.5 million people in the United States. Pressure injuries are classified into four escalating stages, from intact skin to full thickness wounds with deep tissue loss and exposed bone. This study will compare current standard of care treatment (as recommended by the National Pressure Injury Advisory Panel) to treatment with Altrazeal® in patients with stage 2, stage 3 and stage 4 pressure injury wounds. Altrazeal® is a Class 1, 501(k) exempt medical device listed with the FDA as a "dressing, wound, hydrogel" and has an extended wear time of up to 30 days. Subjects can be enrolled in the study either as an outpatient, or while hospitalized. Half of the subjects will be randomized to standard of care treatment, and the other half will be randomized to Altrazeal®. There are a total of up to 12 study visits taking place over 12 weeks.

DETAILED DESCRIPTION:
Pressure injuries, commonly known as pressure ulcers, affect over 2.5 million people in the United States. Pressure injuries are classified into four escalating stages, from intact skin with redness to full thickness wounds with deep tissue loss and exposed bone.

This study will focus on patients with stage 2, stage 3 and stage 4 pressure injury wounds. It will compare current standard of care treatment (as recommended by the National Pressure Injury Advisory Panel) to treatment with Altrazeal® Transforming Powder Dressing (TPD). Altrazeal® is a Class 1, 501(k) exempt medical device listed with the FDA as a "dressing, wound, hydrogel" and has an extended wear time of up to 30 days. Altrazeal® is a powder dressing that conforms to the wound, covering and protecting it, shielding the wound from bacteria. Altrazeal® is used in conjunction with a secondary dressing when needed.

The primary aim of the study is to evaluate whether dressing changes can be reduced during treatment of pressure injuries. The study will also compare wound healing between the group receiving Altrazeal® and the group receiving standard of care dressings, as well as complications, pain, quality of life, and overall costs between the two groups.

Subjects will be randomized into 2 groups, standard of care and Altrazeal®. Half of the subjects will receive current standard of care treatment, and the other half will receive treatment with Altrazeal®. This is an open-label study, meaning that both the subject and the treatment provider will know what study group the subject has been randomized to.

The first visit will be the screening visit to ensure patients meet eligibility criteria. Patients can be either an outpatient or hospitalized. Written informed consent will be obtained during this visit. A wound evaluation will be performed, and laboratory work ordered, if not done recently.

Once identified as meeting study criteria, the next visit is Baseline Visit, where randomization will occur and the first treatment will take place. Participants will be evaluated for 12 additional consecutive weeks, receiving wound evaluation, measurements, and getting treatment for the wound. A pain evaluation, quality of life survey related to having a wound, questionnaire regarding additional wound care performed between study visits. Participants will also answer questions regarding how much offloading devices or maneuvers were utilized, medications taken, and if any complications developed related to their wound care.

If the wound is healed prior to 12 weeks, the study will end when the wound is healed. Otherwise, the study will go on for 12 consecutive weeks. At the end of the study, the participant will be asked to complete a Subject Satisfaction Survey, answering questions regarding how the wound dressing worked for them. The surveys should take 5-10 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years of age;
2. Stage 2, 3, or 4 Pressure Injuries;
3. Wound exudate is mild to moderate;
4. No clinically active wound infection (clinical diagnosis);
5. Able and willing to provide written (not proxy) informed consent;
6. Clinically stable, as determined by assessment of medical history, vital signs, physical examination, and laboratory testing prior to enrollment.

Exclusion Criteria:

1. Known allergy or hypersensitivity to TPD or its components;
2. Pressure injuries classified as unstageable, deep tissue pressure injury, or Stage 1;
3. Heavily exudative wounds;
4. Wound infection as defined as the presence of a least two of the following: local swelling or in duration, erythema >0.5cm around the ulcer in any direction, local tenderness or pain local warmth and purulent discharge;
5. Poorly controlled diabetes with HgbA1C >12 (as documented in the last 3 months);
6. Body Mass Index (BMI) >45 kg/m2;
7. Venous stasis disease or lymphedema in the affected limb (if wound is located on the limb);
8. Moderate to severe chronic limb ischemia Ankle Brachial Index (ABI) <0.7 on the affected limb, if wound is located on the limb);
9. Received immunosuppression or biologics in the last six weeks and/or is expected to receive either at any point during the study;
10. Selected concurrent treatments (e.g., hyperbaric oxygen, topical oxygen therapy, electrical stimulation, ultrasound, cellular or acellular skin substitutes) during study period that may impact study outcomes;
11. Wounds with necrosis unable to undergo prior definitive debridement;
12. Fistulas;
13. Active gangrene;
14. Untreated HIV;
15. Currently pregnant or lactating;
16. Impending organ transplant;
17. Vulnerable populations including prisoners, pediatrics, cognitively impaired, unconscious, and illiterate patients;
18. Unwilling or unable to comply with offloading recommendations;
19. If, in the opinion of the clinical investigator, a subject is a poor candidate for this study because:

    1. Unable to keep research appointments;
    2. Poorly controlled incontinence which may impact study outcomes (e.g., depending on the location of the wound);
    3. Participated in another investigative study within 3 months of enrollment that could interfere with study outcomes;
    4. Active alcohol or substance abuse (cocaine, heroin, or other substances) that may interfere with healing or subject compliance with visit schedules;
    5. Concurrent clinical condition(s) that could pose a health risk to patient or influence outcome of study;
    6. Not suitable for study participation. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of wound dressing changes | 12 weeks
  The number of primary dressing changes for each treatment group will be compared.

SECONDARY OUTCOMES:
Wound healing | 12 weeks
  Wound healing will be measured by using a ruler each week to report length and width of the wound. Percentage of wound area reduction will be calculated for each treatment group and compared.
Complications (problems) from treating the pressure wound | 12 weeks
  Subjects will be asked to report, will be questioned and observed (by the researchers) each study visit for any complications, problems or adverse events related to the study wound that they experience, such as maceration around the wound from the drainage, moisture, or dressing. Complications and adverse events will be compared during the course of the study
Pain in the wound and from dressing changes. | 12 weeks
  Subjects with sensation in the area of the wound will be asked to complete a validated visual analogue scale. This is a simple validated test asking the subject to rate their pain on a 0-10 point level, where 10 is the worst and 0 is no pain. Mean and median pain scores will be compared for each treatment group during the course of the study
Wound Quality of Life | 12 weeks
  Mean and median changes in validated Wound Quality of Life scores will be measured between groups during the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Saxe Johathan, MD, Principal Investigator — Altrazeal Life Sciences Inc
Locations (14):
- United States (14):
  - San Diego VA, San Diego, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Northwestern Medicine, Chicago, Illinois
  - Medstar Franklin Square Medical Center, Baltimore, Maryland
  - Medstar Good Samaritan Hospital, Baltimore, Maryland
  - Rutgers New Jersey Medical School, Ambulatory Care Center-Wound Care Clinic, Newark, New Jersey
  - Northwell Health System/Zucker School of Medicine, Lake Success, New York
  - NYU Langone Hospital-Long Island, Mineola, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - Westchester Medical Center, 100 Woods, Road, Taylor Care Pavillion, Valhalla, New York
  - University of Pittsburgh Medical Center (UPMC) Presbyterian, Pittsburgh, Pennsylvania
  - VA North Texas Healthcare System, Dallas, Texas
  - Michael E. DeBakey Houston VAMC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Pressure Ulcer Advisory Panel, National Pressure Injury Advisory Panel and Pan Pacific Pressure Injury Alliance. Prevention and Treatment of Pressure Ulcers/Injuries: Clinical Practice Guideline. The International Guideline. Emily Haesler (ed.). EPUAP/NPIAP/PPPIA: 2019.
- [Background] Mervis JS, Phillips TJ. Pressure ulcers: Pathophysiology, epidemiology, risk factors, and presentation. J Am Acad Dermatol. 2019 Oct;81(4):881-890. doi: 10.1016/j.jaad.2018.12.069. Epub 2019 Jan 18. PMID 30664905
- [Background] Essex HN, Clark M, Sims J, Warriner A, Cullum N. Health-related quality of life in hospital inpatients with pressure ulceration: assessment using generic health-related quality of life measures. Wound Repair Regen. 2009 Nov-Dec;17(6):797-805. doi: 10.1111/j.1524-475X.2009.00544.x. PMID 19903301
- [Background] Sebba Tosta de Souza DM, Veiga DF, Santos ID, Abla LE, Juliano Y, Ferreira LM. Health-Related Quality of Life in Elderly Patients With Pressure Ulcers in Different Care Settings. J Wound Ostomy Continence Nurs. 2015 Jul-Aug;42(4):352-9. doi: 10.1097/WON.0000000000000142. PMID 26135820
- [Background] https://www.ahrq.gov/patient safety/settings/hospital/resource/pressureulcer/tool/pu1.html#:~:text=Cost%3A%20Press ure%20ulcers%20cost%20%249.1,related%20to%20pressure%20ulcers%20annually.
- See also: Altrazeal (Transforming Powder Dressing) product information — http://www.Altrazeal.info